CLINICAL TRIAL: NCT03288805
Title: Prospective Cohort Study of Chronic Diseases in South China
Brief Title: Cohort Study in South China
Status: Active, not recruiting | Type: Observational
Sponsor: Min Xia (Other)
Collaborators: Guangxi Medical University (Other); Hainan Medical College (Other); Guangzhou No.12 People's Hospital (Other Government); Fujian Medical University (Other); The First Affiliated Hospital of Xiamen University (Other); Shenzhen Fifth People's Hospital (Other); Guangzhou Medical University (Other)
Responsible Party: Sponsor-Investigator, Min Xia, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: 2017YFC0907100
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum ,Urine and fecal samples for biochemical tests, biomarker examination and DNA extraction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Healthy Chinese residents from South China will be recruited and followed up for at least 4 years to evaluate the association between climate, diet and lifestyle and risks for the development of chronic diseases. Physical examination, questionnaire survey and biological sample collection will be conducted at baseline and the incidence of chronic diseases will be investigated during follow-up.

DETAILED DESCRIPTION:
110,000 adult Chinese (35 to 74 years old) without chronic diseases and major disability who have been living in South China including Guangdong, Fujian, Guangxi and Hainan for more than 5 years will be recruited. All participants will be prospectively followed up for the incidence of chronic diseases (stroke, coronary heart disease, malignant neoplasms, chronic obstructive pulmonary diseases, diabetes and hypertension) and their risk factors (impaired glucose tolerance and obesity). Information about socio-demographic, diet, lifestyle, psychological status, medical history and current medication will be collected by questionnaires. Physical examinations including height, weight, waist and hip circumferences, blood pressure, fat mass and vital capacity will be conducted. Besides, blood, urine and fecal samples will be collected for further analysis. Annual meteorological data throughout the study period will also be collected. The associations between climate, diet and lifestyle and risks for chronic diseases will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* adult Chinese (35-74 years old) who have been living in South China including Guangdong, Fujian, Guangxi and Hainan provinces for more than 5 years.

Exclusion Criteria:

* any subject diagnosed with stroke, coronary heart disease, malignancy, chronic obstructive pulmonary disease, diabetes and hypertension.
* any subject who suffer from major disability and cannot participate in the study.

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult Chinese (35-74 years old) who have been living in South China including Guangdong, Fujian, Guangxi and Hainan provinces for more than 5 years.
Sampling Method: Non-Probability Sample
Enrollment: 110000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of chronic disease | 4 years
  Incidence of chronic disease, including stroke, coronary heart disease, cancer, chronic obstructive pulmonary disease, diabetes and hypertension

SECONDARY OUTCOMES:
Risk factors for chronic diseases | 4 years
  Incidence of impaired glucose tolerance and obesity

CONTACTS AND LOCATIONS:
Overall Officials: Min Xia, Principal Investigator — School of Public Health,Nutrition and Food Hygiene,Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No